CLINICAL TRIAL: NCT07277348
Title: Analysis of The Outcomes of Therapeutic Photorefractive Keratectomy Combined With Prophylactic Accelerated Cross-Linking (PRK-Plus), for Treatment of Thin Suspicious Cornea: Short-Term Pilot Study
Brief Title: Analysis of The Outcomes of Therapeutic Photorefractive Keratectomy Combined With Prophylactic Accelerated Cross-Linking (PRK-Plus), for Treatment of Thin Suspicious Cornea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Omar Said, professor, Fayoum University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRK PLUS in thin cornea
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Thin Suspicious Cornea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRK PLUS (Experimental): PRK PLUS
  Interventions: Procedure: PRK PLUS
- Follow up group (No Intervention): follow up with pentacam

INTERVENTIONS:
Procedure: PRK PLUS — therapeutic photorefractive keratectomy combined with prophylactic accelerated cross-linking
  Arms: PRK PLUS

SUMMARY:
analyze the outcomes of therapeutic photorefractive keratectomy combined with prophylactic accelerated cross-linking (PRK-Plus), for treatment of thin suspicious cornea

ELIGIBILITY:
Inclusion Criteria:

1. CCT less than 490 microns
2. K mean more than 46 and/or K max more than 47.
3. Astigmatism cylinder >1.5 D.
4. D value of Belin/Ambrósio Module > 1.6
5. inferior- superior asymmetry or bow-tie pattern with skewed radial axes on tangential maps and abnormal changes on (BAD).
6. Asymmetry topography between 2 eyes, even if neither eye"s topographic pattern is in itself decidedly abnormal.
7. Any significant skewed radial axis with or without inferior steepening, or one diopter or more of inferior steepening in some areas but an I-S value of ,1.4,7.
8. young patients with against-the-rule astigmatic patterns.
9. a PTA value 40% if calculated.
10. Abnormal Topographic Patterns
11. K2 reading of corneal back surface less than [-7].
12. D Value of CSTP > 2.5 in Belin/Ambrósio curve
13. We look at values within the central 5 mm circle; the map should be displayed in the BFTE float mode with an estimated area of 8 mm of diameter:

    * Elevation values on the front surface values > +12 μ
    * Elevation values on the back surface values >+15 μ.
    * If there is any isolated island on either front or back surfaces (in the BFS float mode)

Exclusion Criteria:

1. Eyes diagnosed with KC.
2. CCT less than 450 microns

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
visual acuity improvement measured by LogMAR system | 1 year
  visual acuity improvement measured by LogMAR system